CLINICAL TRIAL: NCT06914037
Title: A Phase 1, Open-Label, Single-Arm Study of the Safety, Pharmacokinetics and Efficacy of CHT101 in Subjects With Relapsed or Refractory T or B Cell Hematological Malignancies
Brief Title: A Clinical Study of CHT101 in CD70-Positive Relapsed or Refractory Hematological Malignancies
Acronym: COURAGE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Nanjing Calmhome Cell and Gene Engineering Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT101HIIT-01
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma (CTCL); NHL (Non-Hodgkin Lymphoma)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHT101 (Experimental): CD70 UCAR-T
  Interventions: Drug: CHT101

INTERVENTIONS:
Drug: CHT101 — CD70 UCAR-T

SUMMARY:
Evaluate the Safety, Pharmacokinetics and Efficacy of CHT101 in Subjects With Relapsed or Refractory T or B Cell Hematological Malignancies

DETAILED DESCRIPTION:
3 planned dose cohorts will be evaluated during dose escalation phase. The dose expansion will be initiated after SRC (safety review committee) reviewing available safety, PK and preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Willing and able to provide written informed consent.
2. Aged 18 to 70 years, male or female.
3. Confirmed CD70 positive in tumor tissue by immunohistochemistry (IHC).
4. Only the following subtypes of hematological malignancies with measurable disease will be enrolled:

   1. Peripheral T cell lymphoma (including peripheral T cell lymphoma NOS, angioimmunoblastic T cell lymphoma, anaplastic large cell lymphoma, etc.) who have failed ≥1 line of systemic therapy.
   2. Cutaneous T cell lymphoma (including mycosis fungoides (MF) or Sézary syndrome (SS) [stage ≥IIB with disease involving two or more compartments or single-compartment disease with large-cell transformation]) who have failed ≥2 lines of systemic therapies.
   3. Aggressive B cell lymphoma who are refractory or relapsed post ≥2 lines of systemic therapies which contain anti-CD20 antibody and anthracyclines.
   4. Indolent B cell lymphoma who are refractory or relapsed post ≥2 lines of systemic therapies which contain anti-CD20 antibody.
   5. Chronic lymphocytic leukemia (CLL) who are refractory or relapsed post ≥2 lines of systemic therapies which contain BTK inhibitor and BCL-2 inhibitor.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Estimated life expectancy ≥12 weeks.
7. Female patients of childbearing potential and male patients must agree to use a highly effective method of contraception from signing ICF through 2 years after last CHT101 infusion.

Exclusion Criteria (abbreviated):

1. History or presence of CNS metastasis, or clinically relevant CNS pathology such as seizure, stroke, severe brain injury, etc.
2. History of solid organ transplantation.
3. Prior treatment with CD70-targeting agents.
4. Prior treatment with CAR-T or other cellular/gene therapies.
5. Ongoing bacterial, viral or fungal infection requiring systemic anti-infectives.
6. Active autoimmune disease requiring immunosuppression.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days of first infusion of CHT101
  Safety
Maximum tolerated dose (MTD) | 28 days of first infusion of CHT101
  Tolerability

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  Adverse events post infusion of CHT101 infusion
Objective response rate (ORR) | 2 years
  The proportion of subjects who achieve CR or PR after CHT101 infusion
Duration of response (DOR) | 2 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Progression-free survival (PFS) | 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression or death of any cause, which occurs first
Overall survival (OS) | 2 years
  The period from the first infusion to any cause of death
Pharmacokinetics (PK) | 2 years
  Concentration levels of CHT101
Pharmacodynamics (PD) | 2 years
  Concentration levels of cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No